CLINICAL TRIAL: NCT07003672
Title: Role of Regional Lung Compliance and Dynamic Transpulmonary Driving Pressure in the Liberation Difficulty in Tracheostomized Patients Receiving Prolonged Mechanical Ventilation
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202401042RINB
Record Dates: First submitted 2024-12-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-12

CONDITIONS: Weaning Failure
Keywords: prolonged mechanical ventilation，PMV; chronic critical illness，CCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project focuses on the analysis of the correlation between transpulmonary driving pressure and uneven lung ventilation and regional lung compliance in patients using prolonged mechanical ventilation (PMV), in order to understand the clinical occurrence of failure of the final spontaneous breathing test and inability to breathe. Respiratory physiology impairments in patients successfully discharged from respirators.

DETAILED DESCRIPTION:
This plan outlines a research project focusing on patients with prolonged ventilator use (PMV), an important manifestation of chronic critical illness (CCI) characterized by prolonged ventilator use after acute illness. This research team has sufficient experience in PMV clinical research and observed that even in the standardized process of weaning from the ventilator, the proportion of patients who successfully weaned from the ventilator was still low. Only 57.9% of the patients were successfully weaned from the ventilator, while the others were Transfer to a long-term care facility or face adverse outcomes. This research project aims to identify important respiratory physiology factors that increase the chances of PMV patients being weaned from ventilators and address a key unanswered question. PMV is often the result of CCI and involves complex clinical challenges such as organ dysfunction, dysregulated immune response, and recurrent infections. Patients' responses to disengagement training vary, often requiring individualized strategies. Conventional lung monitoring using electrical impedance imaging (EIT) can be used to quantify regional hyperinflation and collapse at each level. This method is based on pixel-level changes in respiratory system compliance and depends on whether the patient is fixed or Measured driving pressure, airway pressure (Paw), esophageal pressure (Pes) while accounting for assisted ventilation; EIT monitoring to quantify lung overinflation and collapse Use intrathoracic driving pressure (ΔPLdyn) changes to assess lung compliance at the pixel level change. We will use currently available methods, combining EIT and Pes monitoring, to measure ΔPLdyn in PMV patients. It has been shown in the literature that using ΔPLdyn rather than dynamic airway driving pressure to quantify regional lung overinflation and collapse, that is, compliance changes, is physiologically reasonable and clinically feasible. This method may represent a more accurate assessment of regional lung mechanics associated with the lowest inspiratory effort in the assisted ventilation setting. We hope to understand the changes in regional lung ventilation and compliance of PMV patients during the respirator weaning test through a series of clinical respiratory physiology research processes, in order to find ways to improve the patient's chances of weaning off.

ELIGIBILITY:
Inclusion Criteria:

* Post-tracheostomy patients who are transferred to the subacute respiratory care ward of National Taiwan University Hospital must use respirators for at least 14 days;
* Be at least 20 years old;
* The oxygen concentration required when using the respirator does not exceed 50%

Exclusion Criteria:

* The vital signs are unstable or require continuous use of vasopressors;
* Pregnancy;
* Chronic obstructive pulmonary disease or asthma;
* Those who have contraindications to the placement of esophageal pressure balloons, such as abnormal blood coagulation, esophageal varices, and those who have undergone esophageal or gastric surgery in the past six months;
* Those who have contraindications to the use of electrical impedance tomography, such as heart rhythm regulators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This project hopes to conduct research on patients on prolonged ventilator use (PMV). This group is an important manifestation of chronic severe illness and prolonged use of respirators after acute illness.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
SIMV+PSV（Synchronized intermittent mandatory ventilation + pressure support ventilation) | ．up to 16 weeks
  Timing points for measurement in respiratory physiology assessment include: 1) once when the ventilator is reduced to the lowest supported SIMV+PV mode, and once in the first and fourth hours of the four-hour weaning test period (collar mask), for a total of three times. The measurement tools were the EIT measuring instrument (PulmoVista 500, Dräger Medical, Lübeck, Germany) and the IC measuring instrument Engström Carestation (GE Healthcare, Madison, WI, USA) available in the Department of Respiratory Therapy of our hospital. The methods for measuring EIT 62,64 and IC 57 were as described in the literature30. Tubes will also be installed and connected to the instruments provided by the respiratory therapy department. The esophageal pressure measurement tube is an esophageal balloon similar to a nasogastric tube. The esophageal balloon used in this study has two functions of pressure measurement and nasogastric tube (Nutrivent®), which can be placed for 30 days and has the function of

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
This project focuses on analyzing the correlation between transpulmonary driving pressure, lung ventilation heterogeneity and regional lung compliance in patients with prolonged mechanical ventilation (PMV), so as to understand the clinical causes of failure of the final spontaneous breathing test and inability to breathe. Physiological aspects of breathing in patients successfully discharged from hospital off ventilators.
Supporting Information: Study Protocol